CLINICAL TRIAL: NCT04486690
Title: Neuroprotection During Open Heart Surgery Propofol Versus Ketofol
Brief Title: Neuroprotection During Open Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ghada fouad (Other)
Responsible Party: Sponsor-Investigator, ghada fouad, associate professor of anesthesia, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: (MS/16.05.63)
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Open Heart Surgery
Keywords: propofol; ketofol; neuroprotection; open heart surgery
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: 2 groups of patients subjected to open heart surgery : Propofol group: Propofol, dose 0.5-2 mg/kg.
  * Ketofol group: Ketofol,( dose 0.25-1 mg/kg propofol plus 0.25-1 mg/kg ketamine diluted in normal saline with maintained 1:1 ratio between propofol and ketamine. )
Who Masked: Participant, Investigator
Masking Description: - Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol group (Experimental): * Propofol infusion, 25-150mic/kg/min.
  * Fentanyl infusion, 1-2 mcg/kg/h.
  * Atracurium infusion, 3-12 mic/kg/min
  Interventions: Drug: propofol
- ketofol group (Active Comparator): * Ketofol 25-150 mic/kg/min with propofol to ketamine ratio 1:1.
  * Fentanyl infusion, 1-2 mcg/kg/h.
  * Atracurium infusion, 3-12 mic/kg/min
  Interventions: Drug: Ketofol (propofol to ketamine ratio 1:1)

INTERVENTIONS:
Drug: Ketofol (propofol to ketamine ratio 1:1) — * Ketofol 25-150 mic/kg/min with propofol to ketamine ratio 1:1.
  * Fentanyl infusion, 1-2 mcg/kg/h.
  * Atracurium infusion, 3-12 mic/kg/min
  Arms: ketofol group
Drug: propofol — Propofol infusion, 25-150 mcg/kg/min.
  * Fentanyl infusion, 1-2 mcg/kg/h.
  * Atracurium infusion, 3-12 mic/kg/min.
  Other Names: deprivan
  Arms: propofol group

SUMMARY:
Millions of individuals with coronary artery, or valvular heart disease have been given a new chance at life by heart surgery, but the potential for neurological injury is a great risk .Neural complications - including neurocognitive dysfunction and ischemic complications are complications of cardiac surgery that can restrict the improved quality of life.

Propofol is one of the most popular agents used for induction of anesthesia. propofol reduces cerebral blood flow but maintains coupling with cerebral metabolic rate for oxygen and decreases intracranial pressure, allowing optimal intraoperative conditions.

Ketamine is a non-competitive antagonist of NMDA receptors that has well documented neuroprotective effects against ischemic brain injury and glutamate-induced brain injury. ketamine has neuroprotective effects against oxygen-glucose deprivation injury

DETAILED DESCRIPTION:
The aim of the study is to evaluate neuroprotective effect of mixture of propofol and ketamine (ketofol) as compared to propofol after open heart surgery.

Induction;

* Pre-oxygenation with100% O2 for 3 min.
* Morphine 0.1-0.15 mg/kg
* Fentanyl, dose 3-5 mcg/kg.
* hypnotic agent differs for each group:
* Propofol group: Propofol, dose 0.5-2 mg/kg.
* Ketofol group: Ketofol,( dose 0.25-1 mg/kg propofol plus 0.25-1 mg/kg ketamine diluted in normal saline with maintained 1:1 ratio between propofol and ketamine. )

Catheterization:

1. Central venous catheter: A suitable central venous catheter will be inserted into Right subclavian vein under complete aseptic technique using seldinger technique.
2. Jugular bulb catheterization: Patients is placed in supine position with mild neck extension. The head is placed in neutral position with mild tilt to the opposite side of insertion. Under complete aseptic conditions, the anatomical landmarks for the right internal jugular vein will be identified (at the level of cricoid cartilage, medial to the sternomastoid muscle and lateral to a palpable internal carotid artery). The internal jugular vein will be then cannulated by retrograde insertion of a catheter for sampling of the jugular venous bulb blood. Catheter will be advanced till resistance of the skull base is reached then withdrawn about 1 to 2 mm.

Position of the catheter will be confirmed by antero-posterior and lateral neck C-arm x-ray to verify the correct placement of the catheter tip in the will be sutured to the skin and dressed with sterile gauze

ELIGIBILITY:
Inclusion Criteria:Age between 30 and 70 years of either sex.

* Patients scheduled for elective cardiac surgery using cardiopulmonary bypass (CPB) either valve surgery or coronary artery bypass surgery

Exclusion Criteria:

* Patient refusal.
* Morbidly obese patients.
* Patients with uncontrolled diabetes.
* Patients with pre-existing neurological disease or using anti-psychotics. Severe or uncontrolled renal, hepatic or endocrinal diseases.
* Pregnancy, post-partum or lactating females
* Allergy to one of the agents used.
* Emergency cardiac surgery.
* Re-do surgery.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | from start of surgery and for 24 hours postoperative
  Cerebral oxygenation as indicated by calculation of:
  1. Arterio-Jugular oxygen content difference.
  2. Estimated cerebral metabolic rate for O2(eCMRO2) eCMRO2=Ca- jO2 x(PaCO2 ∕ 100) Where ……. Ca jO2 is arterio-jugular O2 content difference.
     * PaCO2 is arterial CO2 tension

SECONDARY OUTCOMES:
blood pressure measurement | from start of surgery and for 24 hours postoperative
  measurement of invasive blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: mona a hashish, M.D, Study Chair — professor of anesthesia; ahmed m elshamy, master, Principal Investigator — assistant lecturer of anesthesia; ghada f amer, M.D, Principal Investigator — associate professor of anesthesia; magdy m attalaha, M.D, Study Chair — professor of anethesia

IPD SHARING:
Plan to Share IPD: No